CLINICAL TRIAL: NCT06957925
Title: A Cultural-sensitive Act-Belong-Commit-based School Intervention Reduces the Burden of Anxiety and Depression in Adolescents: a Pilot Cluster-randomized Trial From Uganda
Brief Title: ABC School Intervention Among Ugandan Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Davy Vancampfort, Professor, KU Leuven
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUREC 0501-2023
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Depression Disorders
Keywords: act; belong; commit; adolescents; Uganda; anxiety; depression; physical activity; sleep
MeSH Terms: conditions — Anxiety Disorders; Deafness, Autosomal Dominant 20; Depression; Motor Activity

STUDY DESIGN:
Intervention Model Description: pilot cluster-randomized trial
Who Masked: Outcomes Assessor
Masking Description: Masked for group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABC (Experimental)
  Interventions: Behavioral: educational
- Care as usual (No Intervention)

INTERVENTIONS:
Behavioral: educational — Teachers were provided with a manual that could be implemented in a flexible way adapted to the local context of the school consisting of six sessions. The manual assisted teachers to prepare students for success in understanding what is a good mental health (session 1), how to optimize and maintain good mental health, with a particular focus on being mentally, spiritually, socially and physically active including coping with stressors via breathing exercises and progressive muscle relaxation techniques (session 2), physical activity participation (session 3) and sleep hygiene measures (session 4), the importance of belongingness and commitment (session 5), and how to seek support including peer support, community engagement and existing local services (session 6). The first 6 sessions were facilitated by the teacher, and the next 6 by peers.
  Arms: ABC

SUMMARY:
Schools can be pivotal in addressing mental health challenges, especially in low-income settings like Uganda. This pilot cluster-randomized trial examines the impact of a culturally sensitive Act-Belong-Commit (ACT) intervention, combined with physical activity, sleep hygiene and stress management measures on anxiety and depression among Ugandan adolescents attending secondary school. Adolescents from four secondary schools were randomized by school to either a 12-week, weekly two-hour teacher- and peer-led ACT intervention or a care-as-usual control. Anxiety (GAD-7) and depression (PHQ-9-A) were measured at baseline and immediately post-intervention. Childhood trauma (CTQ-SF), self-reported health, wealth, and food security were assessed at baseline. Linear mixed modeling was used to evaluate intervention effects.

DETAILED DESCRIPTION:
Introduction: Schools can be pivotal in addressing mental health challenges, especially in low-income settings like Uganda. However, randomized controlled trials tailored to cultural and contextual factors are scarce. This pilot cluster-randomized trial examines the impact of a culturally sensitive Act-Belong-Commit (ACT) intervention, combined with physical activity, sleep hygiene and stress management measures on anxiety and depression among Ugandan adolescents attending secondary school.

Methods: A total of 2,598 adolescents (1,295 intervention; 1,303 control; 1,199 boys [46.1%]; mean age 16.3 ± 1.0 years) from four secondary schools were randomized by school to either a 12-week, weekly two-hour teacher- and peer-led ACT intervention or a care-as-usual control. Anxiety (GAD-7) and depression (PHQ-9-A) were measured at baseline and immediately post-intervention. Childhood trauma (CTQ-SF), self-reported health, wealth, and food security were assessed at baseline. Linear mixed modeling was used to evaluate intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* All students aged 14 to 17 years in the four schools were screened for depression and anxiety using the Patient Health Questionnaire - 9 (PHQ-9) (Spitzer et al., 1999) and Generalized Anxiety Disorder - 7 (GAD-7) (Spitzer et al., 2006) as part of school health screening service embedded within the study.

Exclusion Criteria:

* None

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2598 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire -9 | 2 weeks
Generalized Anxiety Disorder - 7 | 2 weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire -9 | 2 weeks
  Item 9: suicidal ideation

CONTACTS AND LOCATIONS:
Locations (2):
- Uganda (2):
  - School, Gulu
  - School, Masaka

IPD SHARING:
Plan to Share IPD: No